CLINICAL TRIAL: NCT00697398
Title: Repetitive Trans-cranial Magnetic Stimulation of the Motor Cortex in Fibromyalgia: A Prospective Randomized Blinded Placebo-controlled Study Evaluating the Clinical Efficiency and the Metabolic Correlate in 18FDG-PET
Brief Title: Repetitive Trans-cranial Magnetic Stimulation of the Motor Cortex in Fibromyalgia: A Study Evaluating the Clinical Efficiency and the Metabolic Correlate in 18FDG-PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-A00084-51; 2008-01
Record Dates: First submitted 2008-06-09; First posted 2008-06-13 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2010-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Sound placebo
  Interventions: Other: Transcranial stimulation
- 2 (Experimental): Sound
  Interventions: Other: Transcranial stimulation

INTERVENTIONS:
Other: Transcranial stimulation — Stimulation to white
  Arms: 1
Other: Transcranial stimulation — Repetitive transcranial magnetic stimulation (rTMS)
  Arms: 2

SUMMARY:
Fibromyalgia (FM) syndrome is a chronic pain condition.Repetitive trans-cranial magnetic stimulation (rTMS) was thus suggested in this indication.

DETAILED DESCRIPTION:
We recently demonstrated that these patients exhibit significant perfusion abnormalities in regions of the brain known to be involved in sensory and affective-attentional dimensions of pain processing. These results, in agreement with previous functional magnetic resonance imaging reports, confirm the hypothesis of central sensitization, which provides the rationale for prescription of centrally acting analgesic agents in patients with severe FM.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient, aged from 18 to 65 years
* Patient presenting a primary fibromyalgia answering the criteria of the ACR
* At present painful patient with a digital echelle of the briefing inventory bread superior or equal to 4/10
* Patient presenting a stable treatment since at least 1 less

Exclusion Criteria:

* Patient minor
* pregnant woman
* women in age to procreate without contraception
* patient deprived of freedom further to a court or administrative order
* patient presenting a secondary fibromyalgia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Analgesic efficiency | 36 months

SECONDARY OUTCOMES:
Additional evaluation of the pain | 36 months
Evaluation of the quality of life | 36 months
Evaluation of the tolerance of the treatment | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Guedj, MD, Principal Investigator — Assistance Publique des hopitaux de Marseille
Locations (1):
- Hôpital de la Timone- Service dCentral de Biophysique et de Médecine Nucléaire, Marseille, France

REFERENCES:
- [Derived] Boyer L, Dousset A, Roussel P, Dossetto N, Cammilleri S, Piano V, Khalfa S, Mundler O, Donnet A, Guedj E. rTMS in fibromyalgia: a randomized trial evaluating QoL and its brain metabolic substrate. Neurology. 2014 Apr 8;82(14):1231-8. doi: 10.1212/WNL.0000000000000280. Epub 2014 Mar 26. PMID 24670891